CLINICAL TRIAL: NCT03032315
Title: Clinical Trial to Compare the Pharmacokinetics of TAH Tablet(80/10/12.5mg) in Comparison to the Co-administration of Telmisartan, Amlodipine and Hydrochlorothiazide in Healthy Male Volunteers
Brief Title: Compare the Pharmacokinetics of TAH(80/10/12.5) Tablet in Comparison to the Co-administration of Telmisartan, Amlodipine and Hydrochlorothiazide in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID-TAH-103
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
MeSH Terms: interventions — Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAH(80/10/12.5) tablet (Experimental): Telmisartan/Amlodipine besylate/Hydrochlorothiazide(80/10/12.5) tablet
  Interventions: Drug: TAH Tablet (Telmisartan80/Amlodipine besylate10/Hydrochlorothiazide12.5)
- Telmisartan+Amlodipine besylate+Hydrochlorothiazide (Active Comparator): coadministration of Telmisartan, Amlodipine besylate and Hydrochlorothiazide
  Interventions: Drug: TWYNSTA(Telmisartan+Amlodipine besylate); Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: TAH Tablet (Telmisartan80/Amlodipine besylate10/Hydrochlorothiazide12.5) — Telmisartan 80.0 mg, Amlodipine besylate 13.87 mg (Amlodipine 10 mg), Hydrochlorothiazide 12.5 mg combination-drug would be administered orally once
  Arms: TAH(80/10/12.5) tablet
Drug: TWYNSTA(Telmisartan+Amlodipine besylate) — TWYNSTA 2 Tab. 40/5mg(Telmisartan 40 mg, Amlodipine besylate 6.935 mg(Amlodipine 5 mg) would be administered orally once
  Arms: Telmisartan+Amlodipine besylate+Hydrochlorothiazide
Drug: Hydrochlorothiazide — Dichlozid 1 Tab.(Hydrochlorothiazide 12.5 mg) would be administered orally once
  Arms: Telmisartan+Amlodipine besylate+Hydrochlorothiazide

SUMMARY:
randomized, open-label, single dose, replicate crossover clinical trial to compare the pharmacokinetics of TAH(80/10/12.5) tablet in comparison to the co-administration of telmisartan, amlodipine and hydrochlorothiazide in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers aged 19 to 55 years
2. body mass index (BMI) of 17.5-30.5kg/m2 and weigh more than 55kg
3. Subject does not have congenital or chronic disease and is without pathologic symptom or finding on medical exam.
4. Subject was determined eligible according to the results of clinical laboratory tests like serum test, hematologic test, blood chemistry test, urine test etc. and vital signs, electrocardiography, physical exam etc. performed during the screening exam. 5) willing and able to provide written informed consent

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
2. A subject with a history of gastrointestinal disease or surgery (except simple appendectomy or repair of hernia), which can influence the absorption of the study drug
3. History of regular alcohol consumption (> 210 g/week) within the 6 months before the screening visit.
4. Subjects who take the medication involved in other clinical trials or bioequivalence tests within three months before the first dose medication characters.
5. Seated systolic blood pressure <100mmHg or ≥ 150 mmHg , or diastolic blood pressure of <600mmHg or ≥ 100mmHg at the screening visit
6. History of alcohol or drug abuse within the 12 months before the screening visit
7. Subjects who treated with metabolizing enzyme inducers or inhibitors such as barbitals within 30days prior to the first dosing.
8. Smoker who smoke more than 20 cigarettes per day
9. Subjects who take ethical the count or over the count medicine within 10days before the first investigational product administration.
10. Blood Subjects who do the whole blood donation within two months or component blood donation within 1month prior to the first dosing.
11. Subjects who can increase risk due to clinical test and administration of drugs or has Severe grade / chronic medical, mental condition or abnormal laboratory result that may interfere with the analysis of test results.
12. Subject with known for hypersensitivity reaction to TWYNSTA TAB or dihydropyridine derivatives
13. Subject with known for hypersensitivity reaction to thiazide diuretics or Sulfonamides
14. Patients with biliary obstructive disorder
15. Patients receiving other drugs that affect RAAS such as Angiotensin Receptor Blocker(ARB), ACE inhibitors or aliskiren
16. Combination with aliskiren in Diabetic patient or moderate to severe renal insufficient subjects (glomerular filtration rate<60mL/min/1.73m2)
17. Patients with severe hepatic impairment
18. Patients with severe aortic stenosis
19. Patients with history of shock
20. Patients with anuria
21. Patients with acute or severe renal failure
22. Patients with hyponatraemia hypokalemia
23. Patients with Addison's disease
24. Patients with hypercalcemia of malignancy
25. Who has Galactose intolerance, LAPP lactose intolerance, glucose-galactose malabsorption or genetic disorders
26. Test subjects who is not willing or unable to comply with guidelines described in this protocol
27. A person who is not determined unsuitable to participate in this test by the researchers

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2016-12-27 (Actual); Study Completion 2016-12-27 (Actual)

PRIMARY OUTCOMES:
AUClast | [Time Frame: Hour 0 (Pre-dose), Hour 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 144(Total 18 points)]
Cmax | [Time Frame: Hour 0 (Pre-dose), Hour 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 144 (Total 18 points)]

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Chonbuk, South Korea

IPD SHARING:
Plan to Share IPD: Undecided